CLINICAL TRIAL: NCT05276518
Title: Effect of Single Layer Versus Double Layer Suturing on Healing of Caesarean Uterine Scar: A Randomized Controlled Trial
Brief Title: Double Vers Single in Cesarean Incision
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Sara AbdelRazek Ramadan Hamad, The principal investigator, Ain Shams Maternity Hospital
Other Study IDs: 3/3
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Cesarean Scar Defect

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- o Group (1): 30 cases who will undergo Two Layer Uterine Closure: o After the delivery the first group will undergo Two Layer Uterine Closure: Double-layer closure of the uterine incision will be performed using unlocked continuous Polyglactin thread sutures(1/0) for both layers, with a large portion of the myometrium and the endometrium included in the first layer. The second layer was a continuous running suture that imbricate the first layer, including serosal and myometrial tissue.
  Interventions: Procedure: Closure of cesarean section incision
- o Group (2): 30 cases who will undergo single layer uterine closure.: The second group will undergo continuous unlocked sutures in a single layer, Uterine closure will begin from one corner of the incision and then the uterine incision wound is closed using Polyglactin thread include endometrium, myometrium and serosa
  Interventions: Procedure: Closure of cesarean section incision

INTERVENTIONS:
Procedure: Closure of cesarean section incision — After the delivery the first group will undergo Two Layer Uterine Closure:
  Double-layer closure of the uterine incision will be performed using unlocked continuous Polyglactin thread sutures(1/0) for both layers, with a large portion of the myometrium and the endometrium included in the first layer. The second layer was a continuous running suture that imbricate the first layer, including serosal and myometrial tissue.
  The second group will undergo continuous unlocked sutures in a single layer, Uterine closure will begin from one corner of the incision and then the uterine incision wound is closed using Polyglactin thread include endometrium, myometrium and serosa.

SUMMARY:
To assess the effect of single versus double layer closure of caesarean scar on the residual myometrium on the short & intermediate term.

DETAILED DESCRIPTION:
Caesarean section is the fetal delivery through an open abdominal incision (laparotomy) and an incision in the uterus (hysterotomy). The first caesarean documented occurred in 1020 AD, and since then, the procedure has evolved tremendously. It is now the most common surgery performed in Egypt, with over 1 million women delivered by caesarean every year. The caesarean delivery rate worldwide rose from 5% in 1970 to 31.9% in 2016 An optimal uterine closure should provide better scar healing. Closure of the uterine incision needs to be considered with regards to benefit and potential harm in order to offer the best available surgical care to women undergoing caesarean section. Surgical suturing technique and mechanical tension affecting the surgical wound are the most important factors related to the incisional integrity, especially for minimizing postoperative caesarean delivery scar defects .

Currently, a low-transverse incision is the preferred method of hysterotomy during caesarean delivery. This incision has traditionally been repaired with a two-layer closure. A two-layer closure usually involves a continuous, unlocking layer of absorbable suture with an addition of adds muscular fold to cover the first layer. Studies showed that women whose uterine incisions have been closed by double-layer following caesarean section experienced greater advantages in terms of residual myometrium thickness, healing ratio (residual myometrium thickness/adjacent myometrium thickness), and dysmenorrhea .

The safe cut off thickness of scar in post LSCS uterus varies from 1.5 to 3.5 mm; the thinning of the site is the cause of worry of dehiscence scar or rupture in next pregnancy. Closure of the uterine incision is a key step in caesarean delivery, correct approximation of the cut margins is not guaranteed .

This may be possibly due to edges getting overlapped; and, after remodelling and the process of the healing, thickness of the site of incision is significantly reduced. There is also a very high possibility of inter surgeon variability. It was felt that if there is a suturing technique which ensures correct approximation of all the layers with nil or minimal possibility of inters operator variability, there will not be any thinning of lower segment caesarean section LSCS site, and scarred uterus repaired in this manner will be able to withstand the stress of labor in future .

A growing body of evidence suggests that the surgical technique for uterus closure influences uterine scar defect, but there is still no consensus about optimal uterus closure. Some techniques seem to have the potential to decrease the risk of short-term complications, while others have long-term benefits, such as reduced risk of uterine rupture. Some maternal symptoms are related to the appearance of the uterine scar, and more specifically to a niche in the caesarean scar as a surrogate marker. niche is defined as an indentation in the myometrium of ≥2 mm in depth and is detectable by transvaginal ultrasound (TVUS), preferably with contrast to limit false negatives. Complications in subsequent pregnancies, including uterine rupture and placenta accreta spectrum disorders, are associated with thin residual myometrium .

Many variations in CS technique have been studied. For example, single-layer unlocked uterine incision closure has been compared to double-layer unlocked uterine incision closure. Double layer locked closure has compared to single-layer locked closure, Fear of scar rupture is one of risks involved in a post caesarean pregnancy .

This had led to an increased rate of repeat caesarean delivery in today's times. Closure of the uterine incision is a key step in caesarean section, and it is imperative that an optimal surgical technique be employed for closing a uterine scar. This technique should be able to withstand the stress of subsequent labor. In the existing techniques of uterine closure, single or double layer, correct approximation of the cut margins, that is, decidua-to-decidua, myometrium to myometrium, serosa to serosa is not guaranteed. Also, there are high chances of inter surgeon variability. It was felt that if a suturing technique which ensures correct approximation of all the layers mentioned above with nil or minimal possibility of inter operator variability existed, there will not be any thinning of lower segment caesarean section (LSCS). Further, a scarred uterus repaired in this manner will be able to withstand the stress of labor in future .

To assess the healing of scar and the risk of uterine rupture and other complication, ultrasonography is used in the evaluation of uterine scar 6 weeks after delivery. It has generally been found that, the thicker the uterine scar, the lower the rate of complications. This may be due to that the thicker scar is stronger, and thus performs better than a thinner one .

ELIGIBILITY:
* Inclusion Criteria:

  * Singleton pregnancy.
  * Gestational age between 37 completed weeks to 42 weeks.
  * Patients undergoing elective primary caesarean section.
* Exclusion Criteria:

  * Pregnant women who declined to participate.
  * History of uterine surgery (e.g. hysterotomy, myomectomy, perforation, caesarean section).
  * Presence of maternal disease (diabetes mellitus, connective tissue disorders, uterine malformations).
  * Women Diagnosed with Placenta Accreta Spectrum during the current pregnancy
  * Multiple pregnancy.
  * Chorioamnionitis.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Randomization will be done using computer generated random sequence. Study population will be randomized into one of the two groups:
  * Group (1): 30 cases who will undergo Two Layer Uterine Closure (A)
  * Group (2): 30 cases who will undergo single layer uterine closure (B)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
The residual myometrial thickness at 3 months by trans vaginal us. | 3 months
  Evaluation of the residual myometrial thickness at 3 months after the caesarean section by trans vaginal ultrasonography saline infusion sonohystrography will be done ( in a full bladder patients , Casco speculum will be inserted into vagina followed by insertion of soft non balloon tip catheter 5 French into uterus through vagina then cervix. The speculum was extracted to insert the transducer, 5-10 cc of saline was inserted through the catheter into the uterine cavity to allow the lining of the uterus to be imaged clearly on the ultrasound screen and showed any endometrial abnormality,. Residual myometrial thickness "RMT" is the distance between the tip of the hypo echoic triangle and the surface of anterior uterine wall measured by mm.)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hamed, Asst . Prof, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Sara abdelrazik Ramadan hamad, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No